CLINICAL TRIAL: NCT03379194
Title: Routine Antibiotic Prescription and Resistance Monitoring in Primary Care Physicians: A Nationwide Pragmatic Randomized Controlled Trial
Brief Title: Routine Antibiotic Prescription Monitoring in Primary Care Physicians: A Nationwide Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Bern (Other); University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CEB-NFP72
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Acute Respiratory Tract Infection; Urinary Tract Infections
Keywords: antibiotic prescriptions; resistance; feedback; primary care
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For final data analysis the biostatistician will be blinded for treatment allocation of physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Antibiotic stewardship program' (Experimental): Physicians receive quarterly over 24 months, first in January 2018 postal mail a feedback on their antibiotic prescriptions and updated antibiotic resistance information from the community. With the first letter, educational material, evidence-based guidelines for conditions leading to most outpatient prescriptions in primary care and leaflets for on using antibiotics wisely are provided. Additional material is made available on a study website that can be accessed by each physician in the intervention group by an unique access code.
  Interventions: Behavioral: Antibiotic stewardship program
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Antibiotic stewardship program — Routine feedback on antibiotic prescriptions in addition to evidence based guidelines for the management of acute respiratory and urinary tract infection and patient leaflets for using antibiotics wisely
  Arms: 'Antibiotic stewardship program'

SUMMARY:
Antibiotic resistance is an increasingly serious problem in Switzerland which is associated with the exposure and overall uptake of antibiotics in a population. Reduced antibiotic prescribing for outpatients is paralleled by a decrease in antibiotic resistance rates.

In a recent pragmatic trial, the investigators found only promising yet not very conclusive results as those were present only in some groups. This nationwide antibiotic stewardship program with routine feedback on antibiotic prescribing was not associated with an overall change in antibiotic use. In older children, adolescents, and younger adults fewer antibiotics were prescribed, but not consistently over the entire intervention period.

Hence, the investigators now aim to evaluate a better-tailored program to obtain a better understanding of the effects on patient-relevant outcomes, antibiotic resistance, and the underlying mechanisms leading to different effects in certain subgroups of patients.

The investigators plan to evaluate a nationwide antibiotic stewardship program combining routine prescription feedback with the provision of physician and patient education material for primary care physicians in Switzerland. The project is conducted within the framework of the National Program on antimicrobial resistance by the Swiss National Science Foundation. Also, additional subprojects will be done where we will assess the impact of COVID-19 on AB prescription by comparing the years 2017,2018, and 2019 with the year 2020 data.

DETAILED DESCRIPTION:
This is a randomized pragmatic controlled trial in all primary care physicians in Switzerland e.g. the top 75% antibiotic prescribers. The trial is based on routinely collected individual reimbursement claims data of the three largest Swiss health insurers covering an estimated number of 3.8 million Swiss residents, and on routinely collected surveillance data on antibiotic resistance. A pragmatic trial design is used. Physicians in the intervention group will not have to provide informed consent but they may opt out and decline receiving any interventional information. Physicians in the control group will not be notified. This approach is justifiable and has previously been approved by all Swiss ethical committees. Investigators will take any measures to guarantee the confidentiality of all collected data. Data provided by health insurers on physicians and patients will be completely anonymized.

This is a nationwide study enrolling all registered primary care physicians (general internal medicine and pediatrics) with more than 100 patient contacts in the year prior to the start of the trial. All primary care providers with shared ZSR (Zahlstellenregister) numbers (e.g. ambulatory settings in hospitals where individual physicians cannot be identified) and with less than 100 patient contacts per year will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians in Switzerland board certified with FMH (Foederatio Medicorum Helveticorum) title in general internal medicine or paediatrics & adolescent medicine, above the 25th percentile of antibiotic prescribing, consulting with at least 100 patients per year and with individual Zahlstellenregister number.

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3426 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall antibiotic use | from month 13 to month 24 post randomization (longer term intervention effect).
  Change in prescribed antibiotics per 100 consultations

SECONDARY OUTCOMES:
Overall antibiotic use | from month 1 to 12 post randomization (short-term intervention effect)
  Change in prescribed antibiotics per 100 patient consultations
Overall antibiotic use | from month 1 to month 24 post randomization, with two repeated measurements, over the first and the second 12 month period
  Change in prescribed antibiotics per 100 patient consultations
Use of broad spectrum antibiotics | from month 1 to month 12, and from month 13 to month 24).
  Change in broad spectrum antibiotics use per 100 consultations
  1. quinolones
  2. oral cephalosporines
Hospitalizations rates | from month 1 to month 12, and from month 13 to month 24
  Hospitalizations rates
  1. all-cause
  2. related to infections (DRG-based definition)
Antibiotic use in four specific age groups | from month 1 to month 12, and from month 13 to month 24.
  Antibiotic use per 100 consultations in four specific age groups, in patients
  1. <6 years
  2. 6 to <18 years
  3. 18 to <65 years
  4. ≥ 65 years

CONTACTS AND LOCATIONS:
Overall Officials: Heiner C Bucher, Prof. Dr., Principal Investigator — University Hospital Basel CEB
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aghlmandi S, Halbeisen FS, Saccilotto R, Godet P, Signorell A, Sigrist S, Glinz D, Moffa G, Zeller A, Widmer AF, Kronenberg A, Bielicki J, Bucher HC. Effect of Antibiotic Prescription Audit and Feedback on Antibiotic Prescribing in Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2023 Mar 1;183(3):213-220. doi: 10.1001/jamainternmed.2022.6529. PMID 36745412